CLINICAL TRIAL: NCT01205464
Title: Immunomodulatory and Clinical Effects of Doxycycline on Persistent Symptoms After Treatment of Neuroborreliosis: A Double-blind, Randomised, Crossover Study
Brief Title: Effects of Doxycycline on Persistent Symptoms Post-neuroborreliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Pia Forsberg, Dep. of Infectious Diseases, Faculty of Health Scienses, Linköping University, Sweden
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 151:2004/25331
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2005-02

CONDITIONS: Fatigue; Radicular Pain; Cognitive Dysfunction; Paresthesia; Paresis
Keywords: Persistent symptoms; Doxycycline; Placebo; Neuroborreliosis
MeSH Terms: conditions — Fatigue; Cognitive Dysfunction; Paresthesia; Paresis | interventions — Doxycycline; Tetracycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): Treatment with Capsule Doxycycline 200 mg, once daily, for 21 days.
  Interventions: Drug: Doxycycline
- Sugar pill (Placebo Comparator): Capsule Placebo, 200 mg, once daily, for 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline, 100 mg, 2 capsules once daily, 24 hour time interval, 21 days.
  Other Names: Doxyferm; Vibramycin; Tetracycline
  Arms: Doxycycline
Drug: Placebo — Placebo, 100 mg, 2 capsules once daily, 24 hour dosage interval, 21 days.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The aim of this randomised, double-blind crossover study was to determine whether Doxycycline has an impact on the persistent symptoms post-neuroborreliosis, through alterations in the immune response and whether such an effect could influence the clinical outcome.

DETAILED DESCRIPTION:
Persistent symptoms after treatment of neuroborreliosis (NB) are not uncommon. There is currently no evidence for improvement of symptoms after repeated or prolonged antibiotic treatment. However, clinical observations have indicated that some patients improve during treatment with doxycycline (DOX), but regain the symptoms some time after completed treatment. This may be due to an immunomodulatory effect of the drug. The aim of this randomised, double-blind crossover study was to determine whether DOX has an impact on the persistent symptoms through alterations in the immune response and whether such an effect can influence the clinical outcome.

A total of 15 patients from South-East Sweden with previously adequately diagnosed NB with diverse persistent symptoms ≥6months after antibiotic treatment were randomised in a double-blind, crossover fashion to receive either DOX 200 mg or placebo (PBO) once daily for three weeks, followed by a wash-out period of six weeks and a further three-weeks treatment with either DOX 200 mg or PBO once daily for three weeks. The primary outcome measures were improvement of the persistent symptoms and physical and mental health, evaluated using the visual analogue scale (VAS), the 36-item Short-Form General Health Survey (SF-36) and through physical examination with special emphasis on neurologic status at the follow-up visits. Secondary outcome measures were changes in drug-induced antigen-stimulated and unstimulated cytokine responses.

ELIGIBILITY:
Inclusion Criteria:

* a history of adequately diagnosed and treated neuroborreliosis (presence of intrathecal borrelia-antibody production)
* persistence of symptoms (with debut in conjunction with neuroborreliosis) of typical character, such as headache, radiculitis, cognitive dysfunction, fatigue, mood disorders, paresthesia or paresis > 6 months post-treatment of neuroborreliosis

Exclusion Criteria:

* systemic immunosuppression (treatment with corticosteroids, cytostatics etc)
* ongoing infection at inclusion
* allergy against doxycycline
* pregnancy
* breast feeding
* psychiatric disease
* multiple sclerosis
* rheumatoid arthritis
* diabetes mellitus type 1 or II
* inflammatory systemic diseases
* liver ohc kidney dysfunction
* treatment with didanosine, quinapril, antacids
* malignancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Improvement in persistent symptoms | 12 weeks

SECONDARY OUTCOMES:
Changes in cytokine levels in plasma/serum in patients during treatment with DOX/PBO | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pia Forsberg, MD, Principal Investigator — Department of Infectious Diseases, Faculty of Health Sciences, Linköping university, Sweden
Locations (1):
- Clinic for Infectious Diseases, University Hospital, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Sjowall J, Ledel A, Ernerudh J, Ekerfelt C, Forsberg P. Doxycycline-mediated effects on persistent symptoms and systemic cytokine responses post-neuroborreliosis: a randomized, prospective, cross-over study. BMC Infect Dis. 2012 Aug 10;12:186. doi: 10.1186/1471-2334-12-186. PMID 22876748